CLINICAL TRIAL: NCT02176369
Title: Maintenance Metronomic Per OS Navelbine In Advanced NSCLC Patients After Previous Platinum Based Chemotherapy: A Multicenter Randomized Best Supportive Care Controlled Phase II Study - MA.NI.LA. Trial
Brief Title: Maintenance Low Dose Oral Navelbine In Patients With Non Small Cell Lung Cancer - MA.NI.LA Trial
Acronym: ONC-MANILA12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Regione Lombardia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-MANILA12; 2012-001103-21 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-06-27 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV
Keywords: Non small cell lung cancer (NSCLC); Lung tumor in advanced phase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vinorelbine (Experimental): 50 mg three times a week for a three weeks cycle
  Interventions: Drug: Vinorelbine
- Close observation/Best Supportive Care (No Intervention): Close observation/Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Vinorelbine — Capsule soft (20/30 mg) - 50 mg three times a week (monday, wednesday and friday) for a three weeks cycle (then recycled the next week at the same doses)Treatment will be continued until progression, unacceptable toxicity or death.
  Other Names: Navelbine
  Arms: vinorelbine

SUMMARY:
Non Small Cell Lung Cancer (NSCLC) represents the first cancer related cause of death worldwide with 1.4 millions of deaths every years. Current standard therapies include platinum-containing drugs but at one year from diagnosis the survival rate is still low (30-40%) .

The purpose of this study is to evaluate the role of a platinum-free drug, named Vinorelbine, administered by the so called "metronomic schedule" in order to prolong the progression free survival of patients.

DETAILED DESCRIPTION:
Systemic therapy remains the mainstay of treatment of advanced stage NSCLC. Combination chemotherapy with a platinum-based regimen has emerged as standard therapy for patients with advanced stage disease. Observations supported by the findings of several clinical trial, established the notion that an efficacy plateau had been reached in advanced stage NSCLC patients treated with platinum-containing drugs.

Recent phase III trials suggest the benefit of "switch" and "continuing" maintenance treatment with different drugs. As "switched therapy", Vinorelbine has been selected on the base of its anti-mitotic role. In fact, the use of anti-mitotic drugs at lower dose but with higher frequency (metronomic schedule) seems to augment the anti-angiogenetic effect of this kind of drugs, thus augmenting the efficacy of the therapy.

Therefore, the purpose of the current study is to evaluate the role of a "switched maintenance" with oral vinorelbine administered as a metronomic schedule in terms of Progression Free Survival (PFS) in advanced NSCLC patients with stable disease after first line platinum based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated approved ICF
2. Histologically or cytologically confirmed diagnosis NSCLC diagnosis
3. Stage IV (using AJCC 7th edition, or wet IIIb / IV using the 6th edition), or recurrent locally advanced disease not amenable to radiation or surgery with curative intent and not amenable to concurrent chemoradiation
4. Patients with stable disease, after four-six cycles of platinum-based chemotherapy as first line therapy. Patients with partial or complete response during first line chemotherapy according to RECIST criteria can be enrolled provided that they have stable disease at the study entry.
5. Patients who may have received adjuvant treatment (containing also vinorelbine) at least 6 mos before study entry
6. ECOG performance status 0-2
7. Adequate bone marrow reserve as measured by ANC ≥ 1500/mm3, hemoglobin ≥ 9 g/dL, platelet count ≥ 100,000/μL, ≥ 1 week after last transfusion of blood products and/or last dose of hematopoietic growth factor
8. Prothrombin time (PT) or INR or aPTT ≤ 1.5 x ULN
9. Calculated creatinine clearance ≥ 30 mL/min (Cockcroft and Gault Formula)
10. AST (SGOT) and ALT (SGPT) < 2.5 x ULN, AST and ALT < 5 x ULN (if documented liver metastases)
11. Serum bilirubin < 2.0 mg/dL (patients with Gilbert's syndrome: serum bilirubin ≤ 3 x ULN
12. Alkaline phosphatase < 2.5 x ULN (patients with documented liver or bone metastases, alkaline phosphatase ≤ 5 x ULN)
13. No other obvious related major organ toxicities which would compromise the patient's ability to participate in a clinical trial
14. Allowed prior radiation therapy for local or locally advanced disease providing that any clinically significant adverse effects associated with prior therapy have recovered to Grade 1 or less
15. Women of childbearing potential must have a negative serum pregnancy test and agree to use effective birth control during the trial and for 12 wks after the last treatment dose
16. Males must agree to use effective birth control for themselves or their partner during the trial and for 12 wks after the last treatment dose
17. Life expectancy of at least 12 wks
18. Male or female, age ≥18

Exclusion Criteria:

1. Patients who have received induction therapy with platinum obtaining progressive disease
2. Patients who can benefit from pemetrexed maintenance treatment (adenocarcinoma and ECOG PS 0-1) should be excluded. Enrollment in the trial is permitted for patients who refuse maintenance with pemetrexed or in case of clinical contraindications to pemetrexed therapy (for example renal failure, creatinine clearance ≤ 45 mL/min)
3. Patients who have received, or are scheduled to receive, single agent or combination therapy consisting of chemotherapy, targeted, biological, investigational, hormonal as maintenance treatment
4. Previous treatment for metastatic disease with chemotherapy containing oral or i.v. vinorelbine formulation
5. Last dose of induction chemotherapy < 21 d prior to randomization or > 42 d prior to randomization
6. Concurrent treatment with other experimental drugs.
7. Radiation therapy within 3 wks prior to randomization (palliative radiation therapy is allowed, provided that sites of bone marrow production, i.e., iliac crests are not in the radiation field)
8. Major surgery within 4 wks prior to first study drug administration
9. Active central nervous system (CNS) metastatic disease. Patients with stable CNS disease following completion of radiation therapy and/or surgery are eligible
10. Active or chronically recurrent bleeding (e.g., active peptic ulcer disease)
11. Malabsorption syndrome or any other disorder affecting gastrointestinal absorption
12. Clinically significant infection
13. Clinically significant cardiovascular disease or condition including: congestive heart failure (CHF) requiring therapy, need for anti-arrhythmic therapy for a ventricular arrhythmia, severe conduction disturbance, angina pectoris requiring therapy, medically uncontrolled hypertension per the Investigator's discretion, myocardial infarction within 6 mos prior to first study drug administration, New York Heart Association Class II, III, or IV cardiovascular disease
14. Any other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator
15. History of neoplasm other than curatively treated non-melanoma skin cancer or other carcinoma in situ, that has been resected, unless that prior malignancy was diagnosed and definitely treated at least 3 ys previously with no subsequent evidence of recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Assessed at every 2 cycles (6 wks), 28d after last dose intake and, for patients discontinuing vinolbine for reason other than PD, every 6 wks during Follow Up, up to 18 mos after the enrollment of the Last Patient (LPI)
  PFS: defined as the time from the date of randomization to the date of first documentation of progression, or of death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Assessed at every cycle (3wks), 28d after last dose intake and, during Follow Up, every 3 mos except for patients discontinuing vinolbine for reason other than PD whose assessment is every 6 wks, up to 18 mos after LPI
  OS: defined as the time from the date of randomization to the date of death from any cause or the last date the patient was known to be alive.
Objective Tumor Response Rate (ORR, CR+PR) | Assessed at every 2 cycles (6wks), 28d after last dose intake and, during Follow Up, every 3 mos except for patients discontinuing vinolbine for reason other than PD whose assessment is every 6 wks, up to 18 mos after LPI
  ORR, CR+PR: defined as the proportion of patients with measurable disease at baseline achieving partial or complete overall best response according to RECIST version 1.1 criteria.
Duration of Response (only in patients in CR or PR) | Assessed every two cycles (6wks), 28d after last dose intake and, during Follow Up, every 3 mos except for patients discontinuing vinolbine for reason other than PD whose assessment is every 6 wks, up to 18 mos after LPI
  Duration of Response (only in patients in CR or PR): defined as the time from the date of the first documentation of confirmed objective tumor response to the date of first documentation of objective tumor progression, objective tumor recurrence, or of death due to progressive disease, whichever comes first.
Duration of Post Progression Survival | Assessed at 28d after last dose intake and, during Follow Up, every 3 mos except for patients discontinuing vinolbine for reason other than PD whose assessment is every 6 wks, up to 18 mos after LPI
  Duration of Post Progression Survival: defined as the time from the date of first documentation of objective tumor progression to the date of death from any cause or the last date the patient was known to be alive.
Quality of Life (QoL) according to EORTC QLC30, EORTC QOL-LC13 | Assessed at every 2 cycles (6wks), 28d after last dose intake and, for patients discontinuing vinolbine for reason other than PD, every 6 wks during Follow Up, up to 18 mos after LPI
Overall Safety Profile | Assessed at every cycle (3wks) and 28d after last dose intake up to 18 months after LPI
  Overall Safety Profile, characterized by type, frequency, severity [graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0], timing and relationship to study therapy of adverse events and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Platania, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Alessandro Bertolini, MD, Principal Investigator — A.O. Valtellina e Valchiavenna - Ospedale di Sondrio; Andrea De Monte, Principal Investigator — A.O. Ospedale di Circolo di Melegnano - P.O. Vizzolo Predabissi; Luigi Cavanna, MD, Principal Investigator — AUSL Piacenza - Ospedale Guglielmo da Saliceto; Marco Bregni, MD, Principal Investigator — A.O. Ospedale di Circolo di Busto Arsizio; Yasmina Modena, MD, Principal Investigator — Azienda Ulss18 - Ospedale S.M. della Misericordia - Rovigo; Fabrizio Nelli, MD, Principal Investigator — AUSL Viterbo - Ospedale di Belcolle; Daniele Pozzessere, MD, Principal Investigator — Azienda USL 4 Prato - O.C. Misericordia e Dolce; Hector Soto Parra, MD, Principal Investigator — A. Ospedaliero-Universitaria Policlinico Vittorio Emanuele - Catania; Anna Paola Fraccon, MD, Principal Investigator — Casa di Cura Dott. Pederzoli - Peschiera del Garda; Saverio Cinieri, MD, Principal Investigator — ASL Brindisi - Stabilimento Ospedaliero Di Summa-Perrino; Alessandro Del Conte, MD, Principal Investigator — A.O. Santa Maria Degli Angeli - Pordenone; Vittorio Gebbia, MD, Principal Investigator — Casa di Cura La Maddalena - Palermo; Manlio Mencoboni, MD, Principal Investigator — A.O. Villa Scassi - Genova; Silvia Vattemi, MD, Principal Investigator — ASP di Bolzano - Comprensorio sanitario di Bolzano; Mario Saverio Fumanò, MD, Principal Investigator — Ospedale Morelli - Sondalo; Francesco Verderame, MD, Principal Investigator — A.O.V. Cervello - Palermo; Luciana Irtelli, MD, Principal Investigator — Ospedale Civile SS. Annunziata - Chieti; Graziella Pinotti, MD, Principal Investigator — Ospedale di Circolo e Fondazione Macchi, Varese; Antonio Febbraro, MD, Principal Investigator — Ospedale Sacro Cuore di Gesù Fatebenefratelli - Benevento; Rosa Rita Silva, MD, Principal Investigator — ASUR Marche Area Vasta 2 - Ospedale E. Profili - Fabriano (AN); Gabriella Farina, MD, Principal Investigator — A.O. Fatebenefratelli ed Oftalmico - Milano; Antonio Pazzola, MD, Principal Investigator — Ospedale Civile SS. Annunziata - Sassari
Locations (20):
- Italy (20):
  - Ospedale di Gesù Fatebenefratelli, Benevento, BN
  - ASL Brindisi - Stabilimento Ospedaliero Di Summa-Perrino, Brindisi, BR
  - ASP di Bolzano - Comprensorio sanitario di Bolzano, Bolzano, BZ
  - Ospedale Civile SS. Annunziata, Chieti, CH
  - A. Ospedaliero-Universitaria Policlinico Vittorio Enmanuele, Catania, CT
  - A.O. Villa Scassi, Genova, GE
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - A.O. Ospedale di Circolo di Melegnano - P.O. Vizzolo Predabissi, Vizzolo Predabissi, MI
  - A.O. V. Cervello, Palermo, PA
  - Casa di Cura La Maddalena, Palermo, PA
  - AUSL Piacenza - Ospedale Guglielmo da Saliceto, Piacenza, PC
  - A.O. Santa Maria Degli Angeli, Pordenone, PN
  - Azienda USL 4 Prato - O.C. Misericordia e Dolce, Prato, PO
  - Azienda Ulss18 - Ospedale S.M. della Misericordia, Rovigo, RO
  - Ospedale Morelli, Sondalo, SO
  - A.O. Valtellina e Valchiavenna - Ospedale di Sondrio, Sondrio, SO
  - A.O. Ospedale di Circolo di Busto Arsizio, Busto Arsizio, VA
  - Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Casa di Cura Dott. Pederzoli, Peschiera del Garda, VR
  - AUSL Viterbo - Ospedale di Belcolle, Viterbo, VT